CLINICAL TRIAL: NCT04414098
Title: Safety and Efficacy Study of Ruxolitinib in the Treatment of Severe Acute Respiratory Syndrome Due to SARS-COV-2
Brief Title: Ruxolitinib in the Treatment of Covid-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marcelo Iastrebner (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Marcelo Iastrebner, Principal Investigator, Clinica Zabala
Organization: Clinica Zabala (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZabala
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: Ruxolitinib; Covid-19; SARS
MeSH Terms: conditions — COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Experimental, open-label, prospective, single center, add-on (added to the standard treatment) study, compared with an historical control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: INC424 / Ruxolitinib — 1. Ruxolitinib 5 mg orally every 12 hours during 14 days.
  2. Total Follow-up time will be of 45 days.
  3. The reduction of ruxolitinib dose will be considered in cases of drug-related cytopenias.
  4. During hospitalization, clinical and laboratory evolution parameters will be recorded daily in the medical history of the patient and in the data collection table of the study. Upon patient's discharge, a follow-up will be conducted until day +45
  5. During hospitalization, adverse events will be monitored daily by means of clinical assessment and laboratory data.
  6. After discharge, monitoring of adverse events will continue during the outpatient follow-up.
  7. Pro-inflammatory parameters will be assessed at baseline, after one week (day +7) and at the end of treatment (day +14)
  8. Ruxolitinib will be associated to the standard of care for COVID-19 of each center.
  9. In case of an adverse effect or a need to discontinue the treatment, ruxolitinib should be suspended.
  Other Names: Jakavi

SUMMARY:
The treatment of COVID-19 severe acute respiratory syndrome with ruxolitinib 5 mg orally every 12 hours during 14 days would stop the disproportionate inflammatory response, causing a reduction in the proportion of patients who show a progression and worsening of the severe acute respiratory syndrome.

DETAILED DESCRIPTION:
Primary Objective

Evaluate the efficacy of ruxolitinib in the treatment of COVID-19 severe acute respiratory syndrome by means of measuring the proportion of patients with clinical worsening (defined by a requirement of FIO2 50% and/or mechanical respiratory assistance) during 14 days after the commencement of treatment.

Secondary Objectives

1. Evaluate the median duration of hospitalization. Median duration after 45 days of commencement of treatment.
2. Evaluate the evolution of systemic inflammation parameters. Evaluation at the beginning (baseline), middle and end of the treatment with ruxolitinib of PCR, LDH, ESD, Ferritin and IL-6.
3. Evaluate COVID-19 mortality rate after 45 days of treatment.
4. Evaluate the proportion of the requirement of mechanical ventilation.
5. Evaluate ruxolitinib adverse reactions with a total follow-up of 45 days.
6. Evaluate the proportion of secondary infections during the treatment with ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years.
2. SARS-Cov2 infection confirmed by a validated method.
3. Presence of COVID-19 severe acute respiratory syndrome with:

   Respiratory rate ≥ 20/min O2 saturation ≤93% with FiO2 of 0.21 Lung images by means of computerized tomography or thorax radiography compatible with respiratory involvement due to COVID-19.
4. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or breast-feeding.
2. Platelets < 50,000/mm3.
3. Neutrophils < 1,000/mm3.
4. Hemoglobin < 6 g/dl
5. Creatinine ≥2 mg/dl or creatinine clearance ≤30 ml/min.
6. Total serum bilirubin > 2.0 x upper limit of normal and/or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 times the upper limit of normal.
7. Known active infection due to HIV, HVC, HVB, Herpes Zoster or Micob Tuberculosis
8. Treatment with Tocilizumab, Baricitinib or Interferon.
9. History of hypersensitivity to ruxolitinib or to any medicine with similar chemical compounds
10. Patients with mechanical respiratory assistance
11. Patients under treatment with Ruxolitinib due to hematological disease
12. Any condition that, according to the Investigator, may interfere with the complete participation of the patient in the study, including the administration of the medicinal product, the limitation of visits, the implication of a risk for the patient or that prevents the correct interpretation of the results.

Treatment Suspension Criteria

1. Voluntary decision of the patient
2. Treating physician's decision to discontinue the treatment
3. Drug toxicity grade 3 or higher (CTCAE 5.0).

Study Design

Experimental, open-label, prospective, single center, add-on (added to the standard treatment) study, compared with the historical control arm.

Control arm: It will include patients with COVID-19 Respiratory Syndrome who meet the aforementioned selection criteria and have received the standard of care (SOC). Efforts will be made so that both arms share similar demographic characteristics as regards gender and age group. Ten centers will participate, which will share the same protocol and their results may be jointly analyzed. The expected n per center is 10-15 patients.

For the safety assessment as part of the objective, the following parameters will be taken into account:

1. Biochemical changes: (day 1, 8 and 14) Leukocytes, Formula, Hemoglobin, platelets, creatinine, glycemia, PT, Bilirubin, GOT/GPT.
2. Grade 3/4 Toxicity, SAE (Serious Adverse Event)
3. Incidence of discontinuation, suspension or dose-reduction of the study drug.
4. Incidence of secondary infections.

Efficacy Assessment:

1. Efficacy will be graded according to the ordinal scale of 8 points.
2. Time to Improvement
3. Time of response consolidation
4. Changes in NEWS table

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of ruxolitinib in the treatment of COVID-19 severe acute respiratory syndrome | during 14 days after the commencement of treatment
  Measuring the proportion of patients with clinical worsening (defined by a requirement of FIO2 >50% and/or mechanical respiratory assistance)

SECONDARY OUTCOMES:
Evaluate the median duration of hospitalization. | after 45 days of commencement of treatment.
Evaluate the evolution of systemic inflammation parameters. | after 45 days of commencement of treatment.
  Evaluation at the beginning (baseline), middle and end of the treatment with ruxolitinib of PCR, LDH, ESD, Ferritin and IL-6 (if available).
Evaluate COVID-19 mortality rate | after 45 days of treatment.
Evaluate the proportion of the requirement of mechanical ventilation. | with a total follow-up of 45 days
Evaluate ruxolitinib adverse reactions | with a total follow-up of 45 days.
Evaluate the proportion of secondary infections during the treatment with ruxolitinib | after 45 days of commencement of treatment.

REFERENCES:
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] McGonagle D, Sharif K, O'Regan A, Bridgewood C. The Role of Cytokines including Interleukin-6 in COVID-19 induced Pneumonia and Macrophage Activation Syndrome-Like Disease. Autoimmun Rev. 2020 Jun;19(6):102537. doi: 10.1016/j.autrev.2020.102537. Epub 2020 Apr 3. PMID 32251717
- [Background] Banerjee S, Biehl A, Gadina M, Hasni S, Schwartz DM. JAK-STAT Signaling as a Target for Inflammatory and Autoimmune Diseases: Current and Future Prospects. Drugs. 2017 Apr;77(5):521-546. doi: 10.1007/s40265-017-0701-9. PMID 28255960
- [Background] Zhou Y, Hou Y, Shen J, Huang Y, Martin W, Cheng F. Network-based drug repurposing for novel coronavirus 2019-nCoV/SARS-CoV-2. Cell Discov. 2020 Mar 16;6:14. doi: 10.1038/s41421-020-0153-3. eCollection 2020. PMID 32194980
- [Background] Slostad J, Hoversten P, Haddox CL, Cisak K, Paludo J, Tefferi A. Ruxolitinib as first-line treatment in secondary hemophagocytic lymphohistiocytosis: A single patient experience. Am J Hematol. 2018 Feb;93(2):E47-E49. doi: 10.1002/ajh.24971. Epub 2017 Dec 4. No abstract available. PMID 29134683
- [Background] Harrison CN, Vannucchi AM, Kiladjian JJ, Al-Ali HK, Gisslinger H, Knoops L, Cervantes F, Jones MM, Sun K, McQuitty M, Stalbovskaya V, Gopalakrishna P, Barbui T. Long-term findings from COMFORT-II, a phase 3 study of ruxolitinib vs best available therapy for myelofibrosis. Leukemia. 2016 Aug;30(8):1701-7. doi: 10.1038/leu.2016.148. Epub 2016 May 23. PMID 27211272
- [Background] Gadina M, Le MT, Schwartz DM, Silvennoinen O, Nakayamada S, Yamaoka K, O'Shea JJ. Janus kinases to jakinibs: from basic insights to clinical practice. Rheumatology (Oxford). 2019 Feb 1;58(Suppl 1):i4-i16. doi: 10.1093/rheumatology/key432. PMID 30806710